CLINICAL TRIAL: NCT01606345
Title: Phase I Dose Escalation and Landmark Study of Percutaneous Valrubicin for Upper Tract Urothelial Carcinoma (UTUC) Following Endoscopic Resection
Brief Title: Phase I Study of Percutaneous Valrubicin for Upper Tract Urothelial Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16722
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Urothelial Carcinoma
Keywords: Upper Tract Urothelial Carcinoma; UTUC; Kidney; Cancer; Renal
MeSH Terms: conditions — Carcinoma, Transitional Cell; Neoplasms | interventions — valrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I Dose Escalation (Experimental): Dose escalation: 200 mg/75 ml effluent, 400 mg/75 ml effluent, 800 mg/75 ml effluent
  Interventions: Drug: Valrubicin

INTERVENTIONS:
Drug: Valrubicin — Eligible patients will receive percutaneous valrubicin beginning no sooner than 10 days following nephrostomy placement and within 6 weeks of tumor treatment/resection.
  Other Names: ValstarTM

SUMMARY:
The purpose of this study is to learn more about how well the drug valrubicin (VALSTAR®) works to help treat the patient's cancer when administered through a nephrostomy tube inserted through their back into their kidney. The study is also being done to determine how safe and easy it is to tolerate valrubicin at specific dose levels, as well as the way in which the drug is eliminated from the human body (Pharmacokinetics or PK).

DETAILED DESCRIPTION:
Eligible patients will receive percutaneous valrubicin beginning no sooner than 10 days following nephrostomy placement and within 6 weeks of tumor treatment/resection. Therapy will be administered at one of three dose levels in a 3 + 3 design (200 mg/75 ml diluent, 400 mg/75 ml diluent or 800 mg/75 ml diluent). It is anticipated that at least 3 patients will be accrued at both of the 200 and 400 mg dose levels. Assuming acceptable toxicity, the accrual target for the 800 mg dose level will be 9 patients. If the maximum tolerated dose is determined to be 200 mg or 400 mg, expansion to 9 patients will occur at the maximum tolerated dose (MTD) dose level. Drug will be administered on a weekly basis for 8 total treatments.

ELIGIBILITY:
Inclusion Criteria:

* Zubrod: Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Tissue confirmation of UTUC
* Available tumor grade information
* Treated UTUC (complete resection and or fulguration of tumor as is safely possible, based on the judgment of the investigators and based on visual inspection of the involved kidney and ureter) and at least one of the following:

  * Low grade urothelial carcinoma
  * Percutaneous upper tract Bacillus Calmette-Guérin (BCG) failure and: High grade urothelial carcinoma or Carcinoma in situ (CIS) with imperative indications for nephron preservation (solitary kidney, renal insufficiency, bilateral upper tract tumors, etc.) as determined by study Principal Investigators (PIs)
  * Contraindications to percutaneous BCG (e.g. previous adverse systemic or local reaction to BCG exposure as judged by PIs, or immunosuppression, or other contraindications to BCG therapy) and: High grade urothelial carcinoma or CIS with imperative indications for nephron preservation (solitary kidney, renal insufficiency, bilateral upper tract tumors, etc.) as determined by study PIs
* Normal prothrombin time (PT), partial thromboplastin time (PTT), international normalized ratio (INR)
* Platelets 100 x 10^9/l or greater
* Absolute neutrophil count (ANC) 1.5 x 10^9/l or greater
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) 3 x upper limits of normal (ULN) or less
* Able to receive valrubicin within 6 weeks of the initial surgery or within 6 weeks of a second look surgical procedure

Exclusion Criteria:

* Radiographic or pathologic evidence for locally advanced (muscle invasion, lymphovascular invasion, lymphadenopathy, renal parenchymal invasion) or distant metastatic disease
* Contraindications for percutaneous nephrostomy (i.e. bleeding diathesis and/or patients who must be maintained on therapeutic doses of warfarin or antiplatelet agents while valrubicin is being administered). Note: 81 mg aspirin acceptable.
* Evidence for renal/ureteral obstruction as determined by radiographic studies (antegrade nephrostogram, Intravenous pyelography (IVP), Computed tomography (CT) urogram, retrograde pyelogram, lasix renogram, or a combination thereof)
* Contraindication to percutaneous administration of valrubicin, a metabolite of valrubicin, or known hypersensitivity to anthra-cyclines or polyoxyl castor oil.
* Symptomatic urinary tract infection based on a combination of urinalysis and urine culture and patient symptoms (i.e. Fever). Investigators expect patients to have an abnormal urinalysis based on indwelling urinary devices and prior surgical treatment.
* Urolithiasis in the involved ipsilateral kidney (not including punctuate calcifications or suspected renal parenchymal or papillary tip calcifications seen on radiographic studies or visualized endoscopically)
* Patient on renal replacement therapy (hemodialysis or peritoneal dialysis)
* Extravasation of contrast as visualized on antegrade nephrostogram studies. (Note: At the initial nephrostogram possibly performed in the operating room or with initial percutaneous nephrostomy placement, extravasation can be visualized. However, a procedure prior to drug administration confirms there is not further extravasation present).
* Concurrent malignancy (except basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or concurrent non-muscle invasive bladder cancer that has been completely resected)
* Congenital or acquired immunodeficiency
* Positive pregnancy test or plans for future pregnancy
* Expected poor compliance as judged by the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 12 months
  To define the maximum-tolerated dose (MTD) in a multiple dose regimen of valrubicin administered through a percutaneous nephrostomy tube placed following endoscopic resection (percutaneous or ureteroscopic) of UTUC

SECONDARY OUTCOMES:
Number of Participants with Recurrence Free Survival (RFS) | 12 months
  To evaluate the landmark (1 year) recurrence free survival (RFS). Recurrence is defined as any tumor recurrence in the upper tract following initiation of percutaneous valrubicin.
Number of Participants with Progression Free Survival (PFS) | 12 months
  To evaluate the landmark (1 year) progression free survival (PFS) post valrubicin treatment. Progression is defined as a tumor recurrence in the upper tract of higher clinical stage and/or higher tumor grade following initiation of percutaneous valrubicin.

CONTACTS AND LOCATIONS:
Overall Officials: Wade Sexton, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States